CLINICAL TRIAL: NCT03216083
Title: Does Intravenous Tranexamic Acid Reduce Blood Loss During Vaginectomy? A Double-blind, Placebo-controlled, Randomized Trial
Brief Title: Does Intravenous Tranexamic Acid Reduce Blood Loss During Vaginectomy?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FPMRS McD 002
Record Dates: First submitted 2017-07-10; First posted 2017-07-13 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: colpocleisis; vaginectomy; tranexamic acid
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic Acid (Experimental): Tranexamic Acid Injectable Solution (1g intravenous) Single dose prior to the start of surgery, after the induction of anesthesia
  Interventions: Drug: Tranexamic Acid Injectable Solution
- Placebo (Placebo Comparator): 67mL intravenous normal saline (0.9% sodium chloride) Single dose prior to the start of surgery, after the induction of anesthesia
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid Injectable Solution — 1g IV tranexamic acid mixed in normal saline (67mL)
  Other Names: Cyklokapron
  Arms: Tranexamic Acid
Other: Placebo — 67mL IV normal saline
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
There are many risks for patients undergoing surgery, with blood loss and the risk of resulting anemia and blood transfusion being a common one. Decreasing blood loss with medication can be an important tool in reducing post-operative complications. Tranexamic acid (TXA) is an anti-fibrinolytic that inhibits the activation of plasminogen to plasmin. It inhibits the ability of plasminogen to dissolve fibrin networks, thus decreasing bleeding. TXA was shown in a systematic review and meta-analysis by Ker et. al in 2013 to reduce surgical blood loss by an average of 34% with an increased percentage reduction as the amount of bleeding during surgery decreased. This review also showed that a dose of 1g intravenous (IV) was sufficient in most adults with no evidence supporting a higher dose.

Vaginectomy or total colpocleisis is a surgical procedure performed for women experiencing symptomatic pelvic organ prolapse. It is performed in women who have significant vaginal vault prolapse post-hysterectomy and wish an effective treatment but accept the inability of having penetrative vaginal intercourse. It is most often performed in older patients who have multiple co-morbidities that would preclude them from having a more invasive procedure to correct their prolapse, such as an abdominal sacral colpopexy which involves the placement of surgical mesh, is a significantly longer procedure, and has more associated surgical risks.

This study will be a double-blind, placebo-controlled, randomized trial looking at whether 1g IV tranexamic acid compared with placebo reduces blood loss in women undergoing vaginectomy.

DETAILED DESCRIPTION:
There are many risks for patients undergoing surgery, with blood loss and the risk of resulting anemia and blood transfusion being a common one. Surgeons are constantly working to reduce patient morbidity by decreasing blood loss during procedures. This can be done via excellent surgical technique and meticulous hemostasis but the addition of medications can also be a valuable tool in reducing the amount of blood loss.

Tranexamic acid (TXA) is an anti-fibrinolytic that inhibits the activation of plasminogen to plasmin. It inhibits the ability of plasminogen to dissolve fibrin networks, thus decreasing bleeding. TXA was shown in a systematic review and meta-analysis by Ker et. al in 2013 to reduce surgical blood loss by an average of 34% with an increased percentage reduction as the amount of bleeding during surgery decreased. This review also showed that a dose of 1g intravenous (IV) was sufficient in most adults with no evidence supporting a higher dose.

In gynecology, oral TXA has been used for years in the management of menorrhagia and has been shown to be very effective at decreasing blood loss. In other areas of medicine the IV formulation has shown to reduce death due to bleeding in trauma patients as well as in women experiencing post-partum hemorrhage. Recent RCTs on its use in benign hysterectomy, as well as in advanced ovarian cancer surgery have shown a decrease in blood loss of more than 25% without an increase in adverse events, specifically venous thromboembolic events.

Vaginectomy or total colpocleisis is a surgical procedure performed for women experiencing symptomatic pelvic organ prolapse. It is performed in women who have significant vaginal vault prolapse post-hysterectomy and wish an effective treatment but accept the inability of having penetrative vaginal intercourse. It is most often performed in older patients who have multiple co-morbidities that would preclude them from having a more invasive procedure to correct their prolapse, such as an abdominal sacral colpopexy which involves the placement of surgical mesh, is a significantly longer procedure, and has more associated surgical risks.

Blood loss with a vaginectomy can vary but is not insignificant, especially in elderly women who may have cardiac compromise or pre-existing anemia. The average blood loss quoted in the literature for total colpocleisis varies from 135mL to 396mL, depending on the study. This gives an overall average of about 225mL. If the average patient has a blood volume of 4550mL (calculated based on 65mL/kg in women with a weight of 70kg) this represents a decrease of approximately 5%.

ELIGIBILITY:
Inclusion Criteria:

* female patients over the age of 18
* undergoing a vaginectomy by a member of the Urogynaecology department, with or without concomitant anti-incontinence mid-urethral sling

Exclusion Criteria:

* concomitant hysterectomy at the time of vaginectomy
* inability to read and speak English if no family member or interpreter available for consent process
* cognitively impaired and unable to personally sign consent
* known allergy or intolerance to TXA
* previous venous thromboembolic event
* significant renal impairment (creatinine greater than 200micromol/L or creatinine clearance less than 50mL/min)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin | 4 weeks
  From pre-operative to the morning after surgery

SECONDARY OUTCOMES:
Blood loss | 2 hours
  estimated by surgical team (looking at suction and sponges)
Change in hematocrit | 4 weeks
  From pre-operative to the morning after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Colleen McDermott, MD, Principal Investigator — Mount Sinai Hospital - University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No